CLINICAL TRIAL: NCT06814938
Title: A Novel Precision Medicine Approach for Obesity: a Randomized, Multi-Center Trial
Brief Title: A Study of a Novel Precision Medicine Approach for Obesity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Phenomix Sciences (Unknown)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-006754; 1R44DK138619 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide Group (Experimental): Subjects will take semaglutide weekly for 24 weeks
  Interventions: Drug: Semaglutide
- Placebo Group (Placebo Comparator): Subjects will take placebo weekly for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — 2.4 mg subcutaneous weekly
  Arms: Semaglutide Group
Drug: Placebo — Looks exactly like the study drug, but it contains no active ingredient administered subcutaneous weekly
  Arms: Placebo Group

SUMMARY:
This study is being done to assess the efficacy of a saliva- based biomarker to predict response to semaglutide for the treatment of obesity.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of semaglutide 2.4 mg SQ weekly in patients with obesity with a positive MyPhenome test for abnormal postprandial satiety compared to patients with obesity with a negative MyPhenome test for abnormal postprandial satiety.

ELIGIBILITY:
Inclusion Criteria:

- Obesity (BMI ≥30 kg/m2) without or with controlled chronic conditions (e.g., controlled hypertension).

Exclusion Criteria:

* Weight changes greater than 3% in the previous 3 months
* History of bariatric surgery including lap band and bariatric endoscopy
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD), Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia) and Columbia Suicide Severity Rating Scale (C-SSRS). If such a dysfunction is identified by an anxiety or depression score >11 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up. Any suicidal ideation of type 4 or 5, any suicide attempt during the patient's lifetime, or any suicidal behavior in the last month.
* Current use of anti-obesity medications or GLP1R agonists for Type 2 Diabetes
* Any contraindication to FDA-approved GLP1R agonists
* A person who is pregnant or wanting to become pregnant
* Once the positive or negative cohort is filled at 2:1 ratio, some patients will be screen failed if their gene cohort is full.
* A family member who is enrolled in this study.
* Principal Investigator Discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in Total Body Weight at 24 weeks | Baseline, 24 weeks
  Percent change in body weight in biomarker positive participants vs. biomarker negative participants taking semaglutide vs placebo.

SECONDARY OUTCOMES:
Percentage of Responders >5% | 24 weeks
  Percentage of participants who loss 5% of more of total body weight
Percentage of Responders >10% | 24 weeks
  Percentage of participants who loss 10% of more of total body weight
Percentage of Responders >15% | 24 weeks
  Percentage of participants who loss 15% of more of total body weight
Percentage of Responders >20% | 24 weeks
  Percentage of participants who loss 20% of more of total body weight
Change in Total Body Weight at 3 months | Baseline, 3 months
  Percent change in body weight
Change in Total Body Weight at 6 months | Baseline, 6 months
  Percent change in body weight
Change in Waist Circumference | Baseline, 24 weeks
  Reported in centimeters (CM)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No